CLINICAL TRIAL: NCT06674005
Title: Clinical Trial for the Evaluation of Cucurbita Pepo Flowers Extract to Promote Skin Health
Brief Title: Cucurbita Pepo Flowers Extract to Promote Skin Health
Acronym: EACpLfe22S01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ritamaria Di Lorenzo (Other)
Responsible Party: Sponsor-Investigator, Ritamaria Di Lorenzo, Principal Investigator, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO_CCT22S01; PRO_CCT22S01 (Other: Department of Pharmacy - University of Naples Federico II)
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Skin Laxity; Skin Aging; Skin Wrinkling
Keywords: skin health; wrinkles; collagen; skin resilience
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CpLfe (Active Comparator): Cucurbita pepo L. flower extract at 0.5% w/w in a cosmetic emulgel twice per day for 4 weeks
  Interventions: Other: Cucurbita pepo L. Flowers Extract
- Placebo (Placebo Comparator): cosmetic emulgel twice without the active comparatore twice per day for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cucurbita pepo L. Flowers Extract — 2 mg twice per day for 1 month
  Arms: CpLfe
Other: Placebo — 2 mg twice per day for 1 month
  Arms: Placebo

SUMMARY:
The aim of this cosmetic clinical trial is to learn if an extract of Cucurbita pepo flower (CpLfe) works to enhance skin health and resilience in adult women with photo-damage. It will also learn about the safety of cosmetic active ingredient. The main questions it aims to answer are:

Does cosmetic active ingredient improve skin moisture, luminosity and collagen production, and reduce wrinkles visibility? What skin benefits do participants have when using this new active ingredient in a cosmetic formulation? Researchers will compare the CpLfe to a placebo (a look-alike cosmetic formulation that contains no CpLfe) to see if CpLfe works as ant anti-aging ingredient for skin health.

Participants will:

Take CpLfe or a placebo every day for 1 month Visit the clinic once every 2 weeks for checkups and tests Keep a diary of the potential adverse reactions that might result from using the assigned test products

DETAILED DESCRIPTION:
The skin effects of the CpLfe were evaluated through a double-blind, placebo-controlled, parallel-arm, randomized clinical study. Healthy Italian subjects (age 35-55; n=40) were enrolled in this 4-week study. Before participating, each subject signed a written informed consent that contained the aim and the type of the study, the list of the cosmetic-grade ingredient employed fort the preparation of the cosmetic formulation, the rules to be followed, and any known or potential adverse reactions that might result from using the test products.

All subjects were selected based on the presence of visible wrinkles and skin laxity. Enrolled subjects underwent a 1-week washout period, in which they were instructed to stop using their usual cosmetic products, whereas they were permitted to continue their normal facial treatment regimen (e.g., facial cleanser, make-up removal, eye and lip make-up, and foundation) that did not contain ingredients with anti-aging or lightening action. Once the wash-out period elapsed, subjects were supplied with test products (placebo and the same formulation added with CpLfe).

Panelists had to apply the assigned emulgel twice daily (morning and evening) for 4 weeks. The application amount had to be approximately 0.3 g of product (two pumps) on a dry or slightly moistened face. Massage in, avoiding direct contact with the eyes. Upon application, in case of individual hypersensitivity, discontinue treat-ment. Do not use on irritated or chapped skin. For the evening application wait for at least 1 h before bedtime.

Digital images of all subjects were captured at baseline and at weeks 2 and 4, with VISIA® 7th (Canfield Scientific Inc., Parsippany, NJ 07054 USA). The skin imaging sys-tem exploits IntelliFlash®, cross-polarized light to record and measure skin furrows, folds, and wrinkles. Before image capture, subjects were equilibrated in a controlled temperature room (22 ± 2 °C) for 30 minutes. The hair of the participants was tied up and their clothing was covered with black cloth. The images were taken by the same operator using the same imaging equipment under the same conditions (lighting, dis-tance, head position, etc.) at all time points. Accurate subjects' repositioning was ob-tained by comparing the live image with the ghost-baseline digitally stored photo. Computer analysis of the digital images allowed quantification of the main facial ex-pressive wrinkles (forehead and frown lines, nasolabial folds, and crow's feet).

Facial skin color and spots were also detected through reflectance and spectro-photometric skin devices, like Skin-Colorimeter® CL 400 and Mexameter® MX 18 (Courage+Khazaka electronic GmbH). Specifically, the skin luminosity, melanin index and skin complexion were monitored during the trial. Lastly, facial ultrasonography was carried out, to provide dermis structural organization before and after treatment to confirm the CpLfe ability to firm and densify the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian subjects aged between 35 and 55 y.o.
* Subjects with dull and grey face, lack of firmness, wrinkles, uneven complexion
* Subjects who have read and signed the informed consent
* Subjects who agreed not to apply other products to the test area during the study period
* Subjects who agreed to follow the study procedures and the planned follow-up visits
* Subjects who not change their lifestyle (dermatological and aesthetic medice treatments)
* Absence of systemic pathologies
* Subjects with a good general state of health

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Subjects under 35 and over 55 y.o.
* Subjects with a history of skin hyper-reactivity or intolerance reactions to cosmetic products/ingredients
* Subjects with pathologies in the period immediately preceding the current study
* Subjects undergoing topical or systemic treatment with any drug that may affect the outcome of the test
* Subjects suffering from skin diseases (eczema, psoriasis, lesions)
* Subjects who have undergone dermatological or aesthetic treatments in the six months prior to their recruitment

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
skin hydration | one month
  skin moisture level was measured by Corneometer CM 825 after 2 and 4 weeks of treatment
trans epidermal water loss | one month
  skin trans epidermal water loss was measured with Tewameter TM 300 after 2 and 4 weeks of treatment
collagen production | one month
  dermal collagen was measured with Dermasca C - Probe Ultrasound after 2 and 4 weeks of treatment

SECONDARY OUTCOMES:
Skin luminosity | one month
  skin brightness was measured with Skin-Colorimeter CL 400 (L*-value) after 2 and 4 weeks of treatment
wrinkling | one month
  skin wrinkles were detected through VISIA 7th after 2 and 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Laneri, Professor, Study Director — Federico II University
Locations (1):
- University of Naples Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes
informed consents and results
Supporting Information: Study Protocol, ICF, CSR
Time Frame: one year